CLINICAL TRIAL: NCT04314401
Title: Cancer Moonshot Biobank Research Protocol
Brief Title: National Cancer Institute "Cancer Moonshot Biobank"
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NCI-2020-00750; NCI-2020-00750 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10323 (Other: Division of Cancer Treatment and Diagnosis); 10323 (Other: CTEP)
Record Dates: First submitted 2020-03-18; First posted 2020-03-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Gastric Cancer AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Esophageal Carcinoma; Fallopian Tube Carcinoma; Gastric Carcinoma; Hormone Receptor-Positive Breast Carcinoma; Invasive Breast Carcinoma; Lung Non-Small Cell Carcinoma; Lung Small Cell Carcinoma; Malignant Solid Neoplasm; Melanoma; Metastatic Prostate Carcinoma; Multiple Myeloma; Ovarian Carcinoma; Ovarian High Grade Serous Adenocarcinoma; Primary Peritoneal Carcinoma; Stage III Fallopian Tube Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Esophageal Neoplasms; Fallopian Tube Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Melanoma; Prostatic Neoplasms; Multiple Myeloma; Ovarian Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Triple Negative Breast Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue, bone marrow, cerebral spinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (biospecimen collection, chart review): Patients undergo collection of tissue samples during baseline and at time of disease progression and collection of blood samples throughout the study, including at time of disease progression. Patients with hematological malignancies also undergo collection of bone marrow and cerebral spinal fluid at the same time points. Archival blood and tissue, as well as bone marrow of patients with hematological malignancies, is also collected if available. Additionally, patients may undergo CT, PET/CT and/or MRI throughout the study, and may undergo paracentesis on study. Patient medical records are reviewed, and data is collected for at least 5 years.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Medical Chart Review; Procedure: Paracentesis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, tissue, bone marrow, and cerebral spinal fluid samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Medical Chart Review — Medical charts are reviewed and data is collected
  Other Names: Chart Review
Procedure: Paracentesis — Undergo paracentesis
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT

SUMMARY:
This trial collects multiple tissue and blood samples, along with medical information, from cancer patients. The "Cancer Moonshot Biobank" is a longitudinal study. This means it collects and stores samples and information over time, throughout the course of a patient's cancer treatment. By looking at samples and information collected from the same people over time, researchers hope to better understand how cancer changes over time and over the course of medical treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To support current and future investigations into drug resistance and sensitivity and other National Cancer Institute (NCI)-sponsored cancer research initiatives through the procurement and distribution of multiple longitudinal biospecimens and associated data from a diverse group of cancer patients who are undergoing standard of care treatment at NCI Community Oncology Research Program (NCORP) sites and other National Clinical Trials Network (NCTN) sites.

SECONDARY OBJECTIVES:

I. To provide a service of value to study participants and their medical providers through the performance of molecular profiling assays on tumor samples in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory and reporting of results to physicians and patients that they may opt to use in clinical management, including analysis of data for acquired resistance mechanisms.

II. To enable the development of patient-derived models such as cell lines and xenografts for cancer researchers through the provision of biospecimens from up to 20% of study participants to the NCI's Patient Derived Models Repository (PDMR), a national resource available to investigators.

III. To develop and implement robust approaches in patient and provider engagement to improve understanding of biobanking and its relationship to cancer research and increase representation of minority and underserved study participants in cancer research.

IV. To develop increased capabilities in United States (U.S.) community hospitals and clinics for contribution to cancer research through biobanking activities.

V. To enable secondary research generated from the project through deposition of data in public repositories such as Cancer Research Data Commons (CRDC), The Cancer Imaging Archive (TCIA) and database of Genotypes and Phenotypes (dbGaP) and other potential NCI databases, including clinical, radiology and pathology data with an emphasis on treatment response and outcome data.

VI. To provide residual biospecimens and associated data from the project to the cancer research community.

OUTLINE:

Patients undergo collection of tissue samples during baseline and at time of disease progression and collection of blood samples throughout the study, including at time of disease progression. Patients with hematological malignancies also undergo collection of bone marrow and cerebral spinal fluid at the same time points. Archival blood and tissue, as well as bone marrow of patients with hematological malignancies, is also collected if available. Additionally, patients may undergo computed tomography (CT), positron emission tomography (PET)/CT and/or magnetic resonance imaging (MRI) throughout the study, and may undergo paracentesis on study. Patient medical records are reviewed, and data is collected for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Is consistent with OR has been diagnosed with one of the following:

  * Colorectal cancer: stage IV
  * Non-small cell or small cell lung cancer: stage III/IV
  * Prostate cancer: metastatic prostate cancer
  * Gastric cancer, not otherwise specified (NOS): stage IV
  * Esophageal cancer, NOS: stage IV
  * Adenocarcinoma of gastroesophageal junction: stage IV
  * High grade serous ovarian cancer: stage III/IV
  * Invasive breast carcinoma: stage III/IV
  * Melanoma: stage III/IV
  * Acute myeloid leukemia
  * Multiple myeloma

    * For the purposes of this study,

      * Re-staging is allowed
      * Having more than one primary cancer is allowed, if the patient is being treated solely for one of the eligible cancers listed above
* Patient should fit in one of the following four clinical scenarios (a-d)

  * Undergoing diagnostic workup for one of the diseases listed for which treatment will likely include a new regimen of standard of care therapy OR
  * Scheduled to begin treatment with a new regimen of standard of care therapy OR
  * Currently progressing on a regimen of standard of care therapy OR
  * Currently being treated with a regimen standard of care therapy, without evidence of progression
* Requirements for fresh tissue biospecimen collections at enrollment:

  * For clinical scenarios a, b, and c above, freshly collected tumor tissue or bone marrow (BM) aspirate must be submitted at enrollment

    * For clinical scenarios a and b, the fresh tissue collection must be prior to starting therapy
    * For clinical scenario a, the biospecimen collection must be part of a standard of care medical procedure
    * For clinical scenarios b or c, the biospecimen collection may be part of a standard of care medical procedure OR
    * The biospecimen collection may be part of a study-specific procedure ("research only biopsy"), when the patient has a tumor amenable to image guided or direct vision biopsy and is willing and able to undergo a tumor biopsy for molecular profiling

      * Note: For research-only biopsies, the biopsy must not be associated with a significant risk of severe or major complications or death; the procedure cannot be a mediastinal, laparoscopic, open or endoscopic biopsy; nor can the procedure be a brain biopsy; nor can the patient be under the age of majority as determined by each U.S. state
* Requirements for archival tissue:

  * For clinical scenarios a and b above, archival tissue as outlined below must be submitted IF AVAILABLE
  * For clinical scenarios c and d above, archival tissue as outlined below is REQUIRED
  * Pre-existing archival material (formalin-fixed, paraffin-embedded [FFPE] block, BM aspirate, or unstained slides) that:

    * Contains the cancer type for which the participant is enrolled, and
    * Was collected no more than 5 years prior to initiation of therapy, and
    * Contains at least a surface area of 5 mm^2 and optimal surface area of 25 mm^2 or 3-5 mL cryopreserved bone marrow aspirate to yield 200 million bone marrow mononuclear cells, and
    * Contains at least 10% tumor content. 70% tumor content is optimal, and
    * No more than 1 line of standard of care systemic therapy was administered from the date of archival material collection to the date of initiation of therapy
* Requirements for blood collection: ALL scenarios require fresh blood collection at enrollment

  * Blood collection for clinical scenarios a, b, and c must take place within 1 week of fresh tumor specimen collection
  * Blood collection for clinical scenario d must take place within 4 weeks of enrollment, and while patient is on treatment
* Age 13 or older
* Any sex
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Ability to understand and willingness to sign an informed consent document. Consent may be provided by a Legally Authorized Representative (LAR) in accordance with 45 CFR 46.102(i)
* NCI PDMR INCLUSION CRITERIA: Patients with CRC with mismatch repair deficient (dMMR) or microsatellite instability-high (MSI-H) status
* NCI PDMR INCLUSION CRITERIA: Patients with CRC who are 40 years old or younger at time of collection irrespective of mismatch repair deficient (dMMR) or microsatellite instability-high (MSI-H) status
* NCI PDMR INCLUSION CRITERIA: Patients with BRCA that are either

  * Any race/ethnicity with hormone receptor positive (ER+PR+, ER+PR-, or ER-PR+)
  * African American with triple negative (ER-PR-HER2-)
* NCI PDMR INCLUSION CRITERIA: Patients with lung cancer (LCA), prostate cancer (PCA), gastroesophageal cancer (GEC), ovarian cancer (OV), acute myeloid leukemia (AML), multiple myeloma (MML)

Exclusion Criteria:

* Treated with or has already begun treatment with a non-standard of care therapeutic agent (investigational) in an interventional clinical trial

  * For the purposes of this study, past enrollment in clinical trials whereby the patient was randomized and treated with standard-of-care anti-cancer treatment (chemotherapy regimen, surgery and radiation therapy) is allowed
* Uncontrolled intercurrent illness that in the physician's assessment would pose undue risk for biopsy
* Use of full dose coumarin-derivative anticoagulants such as warfarin are prohibited. Patients may be switched to low molecular weight (LMW) heparin at physician discretion

  * Low molecular weight (LMW) heparin is permitted for prophylactic or therapeutic use
  * Factor X inhibitors are permitted
  * Use of anti-platelet drugs are permitted

    * Stopping the anticoagulation treatment for biopsy, bone marrow aspirate, or resection should be per site standard operating procedure (SOP)
* NCI PDMR EXCLUSION CRITERIA: Patients with complete response
* NCI PDMR EXCLUSION CRITERIA: Patients with invasive fungal infections
* NCI PDMR EXCLUSION CRITERIA: Patients with active and/or uncontrolled infections or who are still recovering from an infection

  * Actively febrile patients with uncertain etiology of febrile episode
  * All antibiotics for non-prophylactic treatment of infection should be completed at least 1 week (7 days) prior to collection
  * No recurrence of fever or other symptoms related to infection for at least 1 week (7 days) following completion of antibiotics
* NCI PDMR EXCLUSION CRITERIA: Patients with human immunodeficiency virus (HIV), active or chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA]) or known history of HBV/HCV without documented resolution

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing treatment for cancer types with commercially available therapies.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-11-11 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Procure, store and distribute longitudinal biospecimens and associated clinical data | Up to 10 years
  Will procure, store and distribute longitudinal biospecimens and associated clinical data for current and future cancer research in order to elucidate molecular mechanisms of sensitivity and intrinsic or acquired resistance to standard of care systemic therapies, including immunotherapy. Cases will be grouped according to patient demographics, cancer type and treatment regimen. Statistical analysis will be descriptive and will be analyzed for each Biospecimen Source Site (BSS) as well as study aggregate.
Percentage of enrolled patients by cancer type and treatment regimen overall | Until completion of biospecimen collection, up to 3 years
  Will assess the percentage of enrolled patients by cancer type and treatment regimen overall and those who contribute samples to the Drug Resistance and Sensitivity Network and other approved investigators. Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate.
Percentage of minority and underserved study participants accrued | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate.

SECONDARY OUTCOMES:
Pan-cancer gene panel tumor next generation sequencing test | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate.
Cancer Research Data Commons, The Cancer Imaging Archive and database of Genotypes and Phenotypes data contribution | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate.
Percentage of minority and underserved study participants accrued | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate.
Percentage of enrolled patients for whom molecular profiling is attempted | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate. Will also be assessed by patient demographics, cancer type and treatment regimen.
Percentage of enrolled patients for whom molecular profiling results are generated | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate. Will also be assessed by patient demographics, cancer type and treatment regimen.
Percentage of enrolled patients for whom samples are obtained at each longitudinal timepoint | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate. Will also be assessed by patient demographics, cancer type and treatment regimen.
Percentage of collected biospecimens that are delivered to the Patient Derived Models Repository | Until completion of biospecimen collection, up to 3 years
  Statistical analysis will be descriptive and will be analyzed for each BSS as well as study aggregate. Will also be assessed by patient demographics, cancer type and treatment regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsay N Harris, Principal Investigator — National Cancer Institute (NCI)
Locations (152):
- United States (149):
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Malbis, Daphne, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Gulf Health Hospitals Inc/Infirmary Cancer Care - Saraland, Saraland, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Veterans Affairs Loma Linda Healthcare System, Loma Linda, California
  - Salinas Valley Memorial, Salinas, California
  - Intermountain Health Platte Valley Hospital, Brighton, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Lutheran Hospital - Cancer Centers of Colorado, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Good Samaritan Hospital - Cancer Centers of Colorado, Lafayette, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - McFarland Clinic - Ames, Ames, Iowa
  - University of Iowa Healthcare Cancer Services Quad Cities, Bettendorf, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Blank Children's Hospital, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Waldo Hospital, Belfast, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Cancer Care and IV Therapy - Brunswick, Brunswick, Maine
  - Mid Coast Hospital, Brunswick, Maine
  - MaineHealth LincolnHealth Hospital, Damariscotta, Maine
  - MaineHealth Franklin Hospital, Farmington, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - MaineHealth Stephens Hospital, Norway, Maine
  - Maine Medical Partners Surgical Care, Portland, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MMP Surgical Care Casco Bay, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Maine Medical Partners Neurology, Scarborough, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - MaineHealth Urology - South Portland, South Portland, Maine
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Newton Medical Center, Newton, New Jersey
  - Chilton Medical Center, Pompton, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Marion L Shepard Cancer Center - ECU Health Beaufort Hospital, Washington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Roger Williams Medical Center, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Baptist Hospital, Columbia, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Monongalia Hospital, Morgantown, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Puerto Rico (3):
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm